CLINICAL TRIAL: NCT05936853
Title: The EPigenetic Consequences in Children of Intravenous vs Volatile Anaesthesia for Surgery (EPIVA) - A Randomised, Feasibility Trial
Brief Title: The EPigenetic Consequences in Children of Intravenous vs Volatile Anaesthesia for Surgery (EPIVA)
Acronym: EPIVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RHM CRI0434
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hypospadias; Anesthesia; Adverse Effect; Perioperative Complication; Pediatric ALL
Keywords: Total intravenous anaesthesia; TIVA; Volatile; Epigenetics; Trial; Surgery; Pediatric; Paediatric; General Anaesthesia
MeSH Terms: conditions — Hypospadias; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to receive maintenance of anaesthesia through either an intravenous approach (TIVA) or inhalational approach (using volatile agents). As is routine anaesthetic practice for this age-group, a gas/inhalational induction will be performed for all participants. After induction a baseline sample of blood will be taken. For participants in the inhalational maintenance group the volatile-based anaesthetic agent (in an air and oxygen mixture) will be continued after induction for the duration of the case. For participants in the TIVA maintenance group, once induction of anaesthesia has been successfully completed, at the earliest appropriate opportunity, the volatile-based anaesthetic will be switched to TIVA which will then be continued for the duration of the case. After the surgical procedure has been completed, and prior to emergence from general anaesthesia, a further blood sample will be taken for analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: It will not be possible to mask the participant's anaesthetist for the case, or the member of the research team. The participant, their Legal Representatives, and the members of the investigation team that are not present for the case, will all remain blinded for the duration of the trial.
  To ensure blinding to arm allocation at the time of outcome analysis/assessment, each participant will also be given a separate 'unique sample identifier code' directly linked to their 'unique participant ID'. This link will not be known by members of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anaesthesia (TIVA) (Active Comparator): This arm will receive maintenance of anaesthesia through a total intravenous anaesthesia approach (TIVA)
  Interventions: Other: Intravenous approach to anaesthetic maintenance
- Inhalational anaesthesia (Active Comparator): This arm will receive maintenance of anaesthesia through an inhalational anaesthesia approach
  Interventions: Other: Inhalational approach to anaesthetic maintenance

INTERVENTIONS:
Other: Intravenous approach to anaesthetic maintenance — Anaesthetic agents given directly into the bloodstream via a cannula.
  Arms: Total intravenous anaesthesia (TIVA)
Other: Inhalational approach to anaesthetic maintenance — Volatile-based anaesthetic drugs are breathed in and then absorbed into the bloodstream through the lungs.
  Arms: Inhalational anaesthesia

SUMMARY:
More than half a million children have an anaesthetic each year in the UK. Though anaesthesia is usually thought to be safe and necessary to improve health, concerns remain the effects that the drugs used may have on brain development in children and the potential long-term consequences for health. The two techniques used to keep someone asleep during anaesthesia are either giving the appropriate drugs through a small plastic tube into a vein or introducing different drugs into the lungs in gas form.

Gene expression is the process by which instructions in DNA are used to make products such as proteins. Anaesthetic drugs may change how a child's genes are expressed; a process called epigenetics. Studies have shown that different anaesthetic drugs can cause epigenetic changes in animals and affect the processing ability of their brains.

This study will focus on children aged under 3 undergoing general anaesthesia for planned hypospadias surgery (a developmental condition where the look and function of the penis may not be completely normally). Participants will either receive their general anaesthetic in gas form or through directly into their veins - both techniques are commonly used. A small blood sample (between 1 and 2 teaspoons) will be collected at the start and end of the operation whilst under anaesthetic. Samples will be analysed to look for any changes in signals on DNA (epigenetic changes) and other markers. Further analysis may then look at other measures of gene expression and additional processes/markers that could be affected.

There is relatively less medical research carried out in children and this work will show whether this type of study is possible in this age-group and provide information for future trials. It will help towards improving our understanding of the effects of anaesthesia ultimately help doctors and families make better informed decisions.

DETAILED DESCRIPTION:
There remains uncertainty about the impact that general anaesthesia may have on many different processes and systems for a child. The effect on the developing brain is an area that has received growing attention over the last decade. Pre-clinical studies, including those looking at cells and animal models, have demonstrated the harmful effect that anaesthetic drugs can cause in nerve cells. Large studies of children have suggested that early age exposure to anaesthetic drugs may impact cognitive and behavioural outcomes however, although this has not been a universal finding.

In 2016 the United States Food and Drug Administration (FDA) issued a warning regarding the use of anaesthetic drugs for children aged under 3 years, with the highest level of concern afforded to those who have prolonged and/or repeat exposures, showing the importance of this topic. This importance is further highlighted by the annual paediatric anaesthetic caseload - more than half a million children have an anaesthetic each year in the UK. There have been pre-clinical studies that have suggested that the way in which anaesthetic drugs can impact on neurodevelopment and cognition is through modifying the way in which genes are expressed by altering signals on DNA (epigenetics). This research aims to explore whether these changes in signals in DNA (epigenetic changes) can be seen in children undergoing anaesthesia and whether this is impacted by the type of anaesthetic given.

To do this, the trial has been designed as a randomised, clinical, feasibility trial in which participants undergoing hypospadias surgery will be randomised to one of the two anaesthetic maintenance approaches that are used routinely in clinical practice: intravenous or inhalational. Baseline data, including demographics, will be collected. On the day of their surgery, participants will receive maintenance of anaesthesia either through inhalational anaesthesia or intravenous anaesthesia according to allocation at randomisation - participants and their legal representatives will be blinded to group allocation and subsequent analysis will be performed with blinding to allocation. The participant will then be anaesthetised, and a baseline blood sample will be taken from the cannula that is routinely inserted into a vein to give medication to the patient. If this is not possible, the sample will be taken from a peripheral site. After the surgical procedure is complete and before the participant wakes up from general anaesthesia, a second blood will be taken. Blood will then undergo laboratory analysis including epigenetic, biochemical, haematological, and redox.

This trial has been designed as a feasibility trial to evaluate whether a larger scale trial looking at anaesthesia and surgery in relation to changes in markers on DNA (epigenetics) is both possible, and of value. Currently there have been no published studies looking at whether general anaesthesia can cause epigenetic changes in children, and whether the type of anaesthetic given has an impact on any changes present. There is significantly less published research in children as it necessitates many additional considerations; this is part of the rationale for this study being designed as a feasibility trial with the primary objective of assessing and determining the feasibility of conducting a paediatric perioperative epigenetics study in which participants are randomised to two methods of maintaining anaesthesia for surgery. Alongside measures such as recruitment and retention rate, screening numbers, protocol compliance figures, this objective will incorporate feedback on acceptability for participants and clinical staff, the success of the data management system used, and if any additional resources are required.

It has also been designed to address the secondary objectives of exploring whether anaesthesia and surgery are associated with epigenetic changes in whole blood, whether the strategy used to maintain anaesthesia impacts any epigenetic changes observed, and to identify which genes, pathways, and functional biological processes, may potentially be involved.

Those with day-to-day responsibility for trial conduct will either be Good Clinical Practice trained trial-team members, or members of the treating clinical team. The Sponsor will continue to have oversight of the trial throughout, and their representatives will communicate closely with the trial team. The end of the study is defined as completion of the full set of analyses of the blood samples taken from participants. The findings will be disseminated in both a timely and responsible manner amongst the relevant scientific community and shared in an appropriate fashion with the legal representatives of the children who took part after. Reporting of the findings may take the form of presentations at meetings/conferences alongside the writing of a manuscript for submission to a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥6 months and ≤ 3 years at time of initial operation
* Undergoing hypospadias surgery
* Maintenance phase of anaesthesia for procedure has an estimated length of ≥1 hour (established through MDT discussion prior to surgery).
* Completed informed consent form (ICF) from legal representative (LR (this is the person who is empowered to give informed consent on behalf of a participant. For most children this will be one or both parents. This may also be a guardian or custodian with legal custody)).

Exclusion Criteria:

* LR unable to provide completed ICF
* Withdrawal of consent at any stage
* Previous exposure to general anaesthesia at any stage of life, including in-utero (through maternal exposure at any stage until delivery)
* Neurodevelopmental/neurodisability diagnosis (given or under investigation) from a paediatric service including autistic specturm disorder (ASD), attention deficit disorder (ADHD), traumatic brain injury (TBI), down's syndrome, cerebral palsy, epilepsy
* Known contraindication to either volatile-based inhalational anaesthesia or TIVA (surgery or participant)
* Clinician refusal

Ages: 6 Months to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of eligible patients screened | 6 months
  Total number of patients during period that would be eligible for the trial
Recruitment rate | 6 months
  Number of participants randomised divided by the number screened
Retention rate | 6 months
  Number of participants that complete the study divided by the number who start it
Protocol compliance | 6 months
  Number of deviations from trial protocol for each patient
Acceptability of trial process for the legal representatives of participants | Up to 1 month
  Outcome to assess whether the legal representatives of participants found the process of partaking in the trial acceptable. This will be self-reported through feedback requests.
Acceptability of trial process for clinical staff | Up to 6 months
  Outcome to assess whether the clinical staff involved in conducting the protocol found this acceptable. This will be self-reported through feedback requests.

SECONDARY OUTCOMES:
Epigenetic changes in whole blood in those undergoing anaesthesia for hypospadias surgery | 5 minutes after induction of anaesthesia, 5 minutes after completion of surgical procedure
  Changes in DNA methylation profile of whole blood (using Illumina Infinium MethylationEPIC BeadChip (850K)) between pre-surgery and post-surgery
Epigenetic changes in whole blood; comparing the two arms of the trial | 5 minutes after induction of anaesthesia and 5 minutes after completion of surgical procedure
  Changes in DNA methylation profile of whole blood (using Illumina Infinium MethylationEPIC BeadChip (850K)) between the two trial arms (TIVA vs inhalational anaesthesia)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Larvin, BMBCH, Principal Investigator — University Hospital Southampton and University of Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available upon request, including the baseline characteristics of patients, feasibility results, and the results of the 850k microarray analysis. Any information is shared and data will remain anonymised at all stages. Age at time of recruitment in years and months will be provided as opposed to date of birth will not be.
  IPD forms part of the informed consent form
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This data will be made available on request from the point of first publication of the results, or 2 years after recruitment is closed.
Access Criteria: Requests for access to the datasets will be discussed by the study's trial management group before any sharing.

REFERENCES:
- [Background] Vutskits L, Xie Z. Lasting impact of general anaesthesia on the brain: mechanisms and relevance. Nat Rev Neurosci. 2016 Oct 18;17(11):705-717. doi: 10.1038/nrn.2016.128. PMID 27752068
- [Background] Vutskits L, Davidson A. Update on developmental anesthesia neurotoxicity. Curr Opin Anaesthesiol. 2017 Jun;30(3):337-342. doi: 10.1097/ACO.0000000000000461. PMID 28277380
- [Background] Jevtovic-Todorovic V, Hartman RE, Izumi Y, Benshoff ND, Dikranian K, Zorumski CF, Olney JW, Wozniak DF. Early exposure to common anesthetic agents causes widespread neurodegeneration in the developing rat brain and persistent learning deficits. J Neurosci. 2003 Feb 1;23(3):876-82. doi: 10.1523/JNEUROSCI.23-03-00876.2003. PMID 12574416
- [Background] Brambrink AM, Back SA, Riddle A, Gong X, Moravec MD, Dissen GA, Creeley CE, Dikranian KT, Olney JW. Isoflurane-induced apoptosis of oligodendrocytes in the neonatal primate brain. Ann Neurol. 2012 Oct;72(4):525-35. doi: 10.1002/ana.23652. PMID 23109147
- [Background] DiMaggio C, Sun LS, Kakavouli A, Byrne MW, Li G. A retrospective cohort study of the association of anesthesia and hernia repair surgery with behavioral and developmental disorders in young children. J Neurosurg Anesthesiol. 2009 Oct;21(4):286-91. doi: 10.1097/ANA.0b013e3181a71f11. PMID 19955889
- [Background] Ing C, DiMaggio C, Whitehouse A, Hegarty MK, Brady J, von Ungern-Sternberg BS, Davidson A, Wood AJ, Li G, Sun LS. Long-term differences in language and cognitive function after childhood exposure to anesthesia. Pediatrics. 2012 Sep;130(3):e476-85. doi: 10.1542/peds.2011-3822. Epub 2012 Aug 20. PMID 22908104
- [Background] Hu D, Flick RP, Zaccariello MJ, Colligan RC, Katusic SK, Schroeder DR, Hanson AC, Buenvenida SL, Gleich SJ, Wilder RT, Sprung J, Warner DO. Association between Exposure of Young Children to Procedures Requiring General Anesthesia and Learning and Behavioral Outcomes in a Population-based Birth Cohort. Anesthesiology. 2017 Aug;127(2):227-240. doi: 10.1097/ALN.0000000000001735. PMID 28609302
- [Background] Warner DO, Zaccariello MJ, Katusic SK, Schroeder DR, Hanson AC, Schulte PJ, Buenvenida SL, Gleich SJ, Wilder RT, Sprung J, Hu D, Voigt RG, Paule MG, Chelonis JJ, Flick RP. Neuropsychological and Behavioral Outcomes after Exposure of Young Children to Procedures Requiring General Anesthesia: The Mayo Anesthesia Safety in Kids (MASK) Study. Anesthesiology. 2018 Jul;129(1):89-105. doi: 10.1097/ALN.0000000000002232. PMID 29672337
- [Background] Ko WR, Huang JY, Chiang YC, Nfor ON, Ko PC, Jan SR, Lung CC, Chang HC, Lin LY, Liaw YP. Risk of autistic disorder after exposure to general anaesthesia and surgery: a nationwide, retrospective matched cohort study. Eur J Anaesthesiol. 2015 May;32(5):303-10. doi: 10.1097/EJA.0000000000000130. PMID 25101714
- [Background] Sun LS, Li G, Miller TL, Salorio C, Byrne MW, Bellinger DC, Ing C, Park R, Radcliffe J, Hays SR, DiMaggio CJ, Cooper TJ, Rauh V, Maxwell LG, Youn A, McGowan FX. Association Between a Single General Anesthesia Exposure Before Age 36 Months and Neurocognitive Outcomes in Later Childhood. JAMA. 2016 Jun 7;315(21):2312-20. doi: 10.1001/jama.2016.6967. PMID 27272582
- [Background] Sury MR, Palmer JH, Cook TM, Pandit JJ. The state of UK anaesthesia: a survey of National Health Service activity in 2013. Br J Anaesth. 2014 Oct;113(4):575-84. doi: 10.1093/bja/aeu292. Epub 2014 Aug 7. PMID 25236896
- [Background] Milanovic D, Pesic V, Loncarevic-Vasiljkovic N, Avramovic V, Tesic V, Jevtovic-Todorovic V, Kanazir S, Ruzdijic S. Neonatal Propofol Anesthesia Changes Expression of Synaptic Plasticity Proteins and Increases Stereotypic and Anxyolitic Behavior in Adult Rats. Neurotox Res. 2017 Aug;32(2):247-263. doi: 10.1007/s12640-017-9730-0. Epub 2017 Apr 24. PMID 28435999
- [Background] Holtkamp C, Koos B, Unterberg M, Rahmel T, Bergmann L, Bazzi Z, Bazzi M, Bukhari H, Adamzik M, Rump K. A novel understanding of postoperative complications: In vitro study of the impact of propofol on epigenetic modifications in cholinergic genes. PLoS One. 2019 May 29;14(5):e0217269. doi: 10.1371/journal.pone.0217269. eCollection 2019. PMID 31141559
- [Background] Bourgeois FT, Murthy S, Pinto C, Olson KL, Ioannidis JP, Mandl KD. Pediatric versus adult drug trials for conditions with high pediatric disease burden. Pediatrics. 2012 Aug;130(2):285-92. doi: 10.1542/peds.2012-0139. Epub 2012 Jul 23. PMID 22826574
- [Background] Joseph PD, Craig JC, Caldwell PH. Clinical trials in children. Br J Clin Pharmacol. 2015 Mar;79(3):357-69. doi: 10.1111/bcp.12305. PMID 24325152
- See also: FDA warning for drugs used for general anaesthesia — https://www.fda.gov/drugs/drug-safety-and-availability/fda-drug-safety-communication-fda-review-results-new-warnings-about-using-general-anesthetics-and